CLINICAL TRIAL: NCT05675137
Title: Efficacy of a Mobile-based Multidomain Intervention to Improve Cognitive Function and Health-related Outcomes Among Older Korean Adults With a High Risk of Dementia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Silvia Health (Industry)
Collaborators: Chosun University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 2022-03-013
Record Dates: First submitted 2022-12-30; First posted 2023-01-09 (Actual); Last update posted 2023-01-09 (Actual); Status verified 2023-01

CONDITIONS: Cognitive Decline; Cognitive Impairment, Mild; Aging; Dementia
MeSH Terms: conditions — Cognitive Dysfunction; Dementia

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mobile-based multidomain intervention (Experimental)
  Interventions: Device: mobile-based
- paper-based intervention group (Active Comparator)
  Interventions: Other: paper-based

INTERVENTIONS:
Device: mobile-based — Participants who were randomly assigned to the mobile-based intervention group were provided multidomain programs based on scientific evidence of ways to improve brain-health and reduce dementia risk for 10 minutes per day and at least 50 minutes per week.
  Arms: Mobile-based multidomain intervention
Other: paper-based — Participants who were randomly assigned to the paper-based intervention group were provided with the Korean version of the dementia prevention booklet published by the WHO.
  Arms: paper-based intervention group

SUMMARY:
This study investigated the efficacy of the Silvia program, a mobile-based multidomain intervention, to improve cognitive function and health-related outcomes of older adults with a high risk of dementia. We compare its effects to a conventional paper-based multidomain program on various health indicators related to risk factors of dementia.

ELIGIBILITY:
Inclusion Criteria:

1. experiencing subjective cognitive decline,
2. had a smart phone and could use it, and
3. understood the purpose and process of this study.

Exclusion Criteria:

1. major psychiatric disorders
2. dementia,
3. degenerative brain diseases
4. severe or unstable heart diseases
5. neurological or psychological diseases that affected cognitive functioning
6. severe vision or hearing impairment,
7. current participation in a cognitive training program
8. does not know how to use mobile devices.

Ages: 60 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2022-04-10 (Actual); Primary Completion 2022-10-28 (Actual); Study Completion 2022-10-28 (Actual)

PRIMARY OUTCOMES:
Change from baseline Korean version of the Repeatable Battery for the Assessment of Neuropsychological status at 12 weeks | baseline and after the 12-week intervention
  Cognitive function

SECONDARY OUTCOMES:
Change from baseline Korean version of the mini-mental state examination, 2nd edition(K-MMSE-2) at 12 weeks | baseline and after the 12-week intervention
  Cognitive function
Change form baseline Korean version of the prospective and retrospective memory questionnaire(K-PRMQ) at 12 weeks | baseline and after the 12-week intervention
  Self-reported memory failures
Change from baseline Center for Epidemiological Studies Depression (CES-D) questionnaire at 12 weeks | baseline and after the 12-week intervention
  Depression
Change from baseline State-Trait Anxiety Inventory-X-1(STAI-X-1) at 12 weeks | baseline and after the 12-week intervention
  Anxiety
Change from baseline Perceived Stress Scale (PSS) at 12 weeks | baseline and after the 12-week intervention
  Stress
Change from baseline EuroQoL 5-Dimension 5-Level(EQ-5D-5L) at 12 weeks | baseline and after the 12-week intervention
  Health-related Quality of life

CONTACTS AND LOCATIONS:
Locations (1):
- Silviahealth, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No